CLINICAL TRIAL: NCT00170664
Title: Taxol/ Carboplatin as First Line Therapy in Patients With Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020114
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian neoplasms; paclitaxel, carboplatin; clinical trials, phase II; first-line chemotherapy; weekly therapy schedule
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin

ARMS (1):
- Paclitaxel, Carboplatin (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The combination of paclitaxel and carboplatin in a three weeks schedule has emerged as the current standard approach for the adjuvant treatment of ovarian cancer. Based on a phase I study now a multi-center phase II-trial was conducted.

ELIGIBILITY:
Inclusion Criteria:

* histologically-confirmed epithelial ovarian cancer of FIGO stage IIB - IV
* life expectancy of more than three months
* ECOG performance status less than 3
* laboratory parameters within the normal range, including a glomerular filtration rate (GFR) greater than 60 ml/min, serum creatinine levels below 1.6 mg/dl, liver transaminases less than two times the normal levels, bilirubin concentrations below 1.5 mg/dl, adequate bone marrow function as indicated by a neutrophil count greater than 1,500/µl, and a platelet count greater than 100,000/µl.
* written informed consent

Exclusion Criteria:

* suffering from secondary malignancy or underlying serious, uncontrolled concurrent medical or psychiatric disease
* radiotherapy within 4 weeks for study entry

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 1999-01; Primary Completion 2003-03 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Lichtenegger, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany